CLINICAL TRIAL: NCT07163754
Title: Use of the SiDTM v2.0 Algorithm to Assist Embryologists in Sperm Selection During ICSI Procedures: Impact in Biological and Clinical Outcomes
Brief Title: Use of the SiDTM v2.0 Algorithm to Assist Embiyologists in Sperm Selection During ICSI Procedures
Acronym: SID_3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: IVF 2.0 Limited (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2502-VLC-027-MM
Record Dates: First submitted 2025-07-17; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Male Fertility; Testicular; Sperm Parameters in Fertile and Infertile Men; Sperm Selection
Keywords: Intracytoplasmatic Sperm injection; automated sperm selection; artificial intelligence; fertilization; embryo quality

STUDY DESIGN:
Intervention Model Description: The present project will be a single-center, open-label, prospective, cohort study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SID (Experimental): Half of the MII oocytes obtained will be microinjected with spermatozoa selected by SiD TM
  Interventions: Diagnostic Test: Automated Sperm Selection
- NO-SID (Active Comparator): Half of the MII oocytes obtained will be microinjected with spermatozoa selected by embriologist.
  Interventions: Diagnostic Test: Conventional Sperm Selection

INTERVENTIONS:
Diagnostic Test: Automated Sperm Selection — This group of oocytes will be microinjected with sperm selected by the second version of SID TM (SID V2.0) wich analyses additional sperm parameters than first version of SID TM (SID V1.0).
  Arms: SID
Diagnostic Test: Conventional Sperm Selection — Half of the oocytes will be microinjected with sperm selected by the embryologist without SID assistance, based on the conventional and visual assesment of seminal samples located at ICSI dishes.
  Arms: NO-SID

SUMMARY:
Infertility is defined as a failure of a couple to achieve a pregnancy after 12 or more months of unprotected intercourse. Males are found to be solely responsible for 20-30% of infertility cases but contribute to 50% of cases overall. The selection of sperm to microinject is completely subjective and there is high intra- and inter- observer variability. SiDTM v2.0 is an algorithm which analyses real-time seminal samples located at ICSI dishes. Particularly, it assesses morphology and several motility parameters of each sperm, and it assigns a categorical and numerical score to each one. Categorical scores are represented by colours: green colour for optimal sperm, yellow for good sperm, orange for medium-quality sperm and red for low-quality sperm. Numerical scores ranged from 0 to 100, with higher scores for those best-quality sperm. SiDTM v2.0 can reduce subjectivity of the sperm selection process to the maximum, selecting the optimal sperm in real time. In addition, it could help junior embryologists to perform this complex and tedious procedure, which is the sperm selection for ICSI. To carry out the study, we will conduct a prospective cohort study in a total of 100 couples. Therefore, the aim of this study is to validate SiDTM v2.0 as an useful Artificial Intelligence-tool for sperm selection; that means achieving , at least, same clinical results as sperm selection performed by the embryologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for ICSI.
* Women of advanced maternal age (>35 years) in whom at least 4 oocytes in metaphase II stages are obtained in the follicular puncture, without excluding patients from the oocyte donation program.
* Sperm obtained by masturbation with a concentration above 1 million spermatozoa/mL after sperm capacitation.
* Normal karyotype of both partners.
* Informed Consent (IC).

Exclusion Criteria:

* Patients diagnosed with recurrent gestational loss.
* Semen extracted by testicular biopsy.
* Semen samples with globozoospermia (sperm defect due to lack of acrosome) or azoospermia (absence of spermatozoa in the ejaculate).
* Semen samples treated with pentoxifylline.
* ICSI cycles with application of calcium ionophore. o ICSI cycles with application of calcium ionophore.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
SID TM V2.0 VALIDATION | 1 year
  The main objective of this study is to test whether assisted sperm selection using the artificial intelligence algorithm SiDTM v2.0 equals or exceeds the mean rate of useful blastocysts obtained by conventional unassisted sperm selection by SiDTM v2.0.

SECONDARY OUTCOMES:
Fertilization assesment (SID vs NO SID) | 1 year
  Fertilization rate (SID VS NO SID)
Embryo development assesment (SID vs NO SID) | 1 year
  Embryo development rate (SID VS NO SID)
Clinical outcomes assesment (SID vs NO SID) | 1 year
  Gestation rate.
Clinical outcomes assesment (SID vs NO SID) | 1 year
  Implantation rate
Clinical outcomes assesment (SID vs NO SID) | 1 year
  Live birth rate.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Meseguer, PhD, Principal Investigator — IVIRMA Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montjean D, Godin Page MH, Pacios C, Calve A, Hamiche G, Benkhalifa M, Miron P. Automated Single-Sperm Selection Software (SiD) during ICSI: A Prospective Sibling Oocyte Evaluation. Med Sci (Basel). 2024 Mar 27;12(2):19. doi: 10.3390/medsci12020019. PMID 38651413
- [Background] Mendizabal-Ruiz G, Chavez-Badiola A, Aguilar Figueroa I, Martinez Nuno V, Flores-Saiffe Farias A, Valencia-Murilloa R, Drakeley A, Garcia-Sandoval JP, Cohen J. Computer software (SiD) assisted real-time single sperm selection associated with fertilization and blastocyst formation. Reprod Biomed Online. 2022 Oct;45(4):703-711. doi: 10.1016/j.rbmo.2022.03.036. Epub 2022 Apr 10. PMID 35989168
- [Background] Carrión-Sisternas, L., Bori, L., Conversa, L., Viloria, T., Tejera, A. AUTOMATED REAL-TIME SPERM SELECTION FOR INTRACYTOPLASMIC SPERM INJECTION (ICSI): SIBLING OOCYTE EVALUATION. Fertility and Sterility, Volume 122, Issue 4, e350
- [Background] Asada Y. Evolution of intracytoplasmic sperm injection: From initial challenges to wider applications. Reprod Med Biol. 2024 May 27;23(1):e12582. doi: 10.1002/rmb2.12582. eCollection 2024 Jan-Dec. PMID 38803410
- See also: Related Info — https://www.ivf20.ai/sid/